CLINICAL TRIAL: NCT00598169
Title: Safety and Efficacy Pilot Trial of the Anti-Viral and Anti-Tumor Activity of Velcade Combined With (R)ICE in Subjects With EBV and/or HHV-8 Positive Relapsed/Refractory AIDS-Associated Non-Hodgkin's Lymphoma
Brief Title: Bortezomib, Ifosfamide, Carboplatin, and Etoposide, With or Without Rituximab, in Treating Patients With Relapsed or Refractory AIDS-Related Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-053; U01CA121947 (NIH); CDR0000581078 (Other: NCI)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Bortezomib; Carboplatin; Dexamethasone; Etoposide; Ifosfamide; Polymerase Chain Reaction; Blotting, Western

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD20+ Non-Hodgkin Lymphoma (Experimental): Part A: Velcade Day 1 and Day 8, with inter-subject dose escalation over four dose levels: 0.7 mg/m2, 1 mg/m2, 1.3 mg/m2 and 1.5 mg/m2. Dexamethasone 20 mg IV and etoposide 100 mg/m2 IV Days 8-10, carboplatin dosed to AUC=5 (maximum 750 mg) IV and ifosfamide 5000 mg/m2 mixed with an equal amount of Mesna on Day 9 of a 28-day cycle.
  Part B: Velcade on Days 1 and 8, dexamethasone 20 mg IV Days 1-3 and Day 8; etoposide 100 mg/m2 IV on Days 1-3; carboplatin dosed to AUC=5 (maximum 750 mg) IV on Day 2; ifosfamide 5000 mg/m2 mixed with an equal amount of Mesna and administered as a continuous IV infusion over 24 hours on Day 2, rituximab 375mg/m2 on Day 1 of a 21-day cycle.
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: carboplatin; Drug: dexamethasone; Drug: etoposide; Drug: ifosfamide; Genetic: polymerase chain reaction; Genetic: western blotting
- CD20- Non-Hodgkin Lymphoma (Experimental): Part A: Velcade Day 1 and Day 8, with inter-subject dose escalation over four dose levels: 0.7 mg/m2, 1 mg/m2, 1.3 mg/m2 and 1.5 mg/m2. Dexamethasone 20 mg IV and etoposide 100 mg/m2 IV Days 8-10, carboplatin dosed to AUC=5 (maximum 750 mg) IV and ifosfamide 5000 mg/m2 mixed with an equal amount of Mesna on Day 9 of a 28-day cycle.
  Part B: Velcade on Days 1 and 8, dexamethasone 20 mg IV Days 1-3 and Day 8; etoposide 100 mg/m2 IV on Days 1-3; carboplatin dosed to AUC=5 (maximum 750 mg) IV on Day 2; ifosfamide 5000 mg/m2 mixed with an equal amount of Mesna and administered as a continuous IV infusion over 24 hours on Day 2, 21-day cycle.
  Interventions: Drug: bortezomib; Drug: carboplatin; Drug: dexamethasone; Drug: etoposide; Drug: ifosfamide; Genetic: polymerase chain reaction; Genetic: western blotting

INTERVENTIONS:
Biological: rituximab — 375mg/m2 on Day 1
  Arms: CD20+ Non-Hodgkin Lymphoma
Drug: bortezomib — Part A: Velcade Day 1 and Day 8 of a 28-day cycle, with inter-subject dose escalation over four dose levels: 0.7 mg/m2, 1 mg/m2, 1.3 mg/m2 and 1.5 mg/m2 Part B: Velcade on Days 1 and 8 of a 21-day cycle.
Drug: carboplatin — Carboplatin will be dosed to an AUC=5, calculated using the Calvert formula (5 x [creatinine clearance + 25]; the maximum dose of carboplatin is 750 mg.
  Part A: AUC=5 (maximum 750 mg) IV administered on Day 9. Part B: AUC=5 (maximum 750 mg) IV administered on Day 2.
Drug: dexamethasone — Part A: 20 mg IV on Days 8-10. Part B: 20 mg IV on Days 1-3 and on Day 8.
Drug: etoposide — Part A: 100 mg/m2 IV Days 8-10. Part B: 100 mg/m2 IV daily on Days 1 to 3.
Drug: ifosfamide — Part A: 5000 mg/m2 mixed with an equal amount of Mesna as a 24 hour continuous IV infusion on Day 9.
  Part B: 5000 mg/m2 mixed with an equal dose of Mesna administered via continuous infusion for 24 hours beginning on Day 2.
Genetic: polymerase chain reaction — Correlate EBV/HHV-8 viral load changes with lymphoma response. HIV and EBV/HHV-8 viral loads will be assessed on baseline, day 2, 4, and 8 of week 1 of Part A.
Genetic: western blotting — Peripheral blood mononuclear cells will be collected at Day 1 prior to chemotherapy, Day 2, 4 and 8 (prior to chemotherapy) then weekly during Part A, just prior to each additional cycle of Part B and at treatment completion. Western blot using antibody specific for APOBEC3G and antibody against actin for internal control will be used to quantify APOBEC3G levels. Changes at will be compared with baseline using a paired t-test.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as dexamethasone, ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving bortezomib together with combination chemotherapy is more effective with or without rituximab in treating AIDS-related non-Hodgkin lymphoma.

PURPOSE: This clinical trial is studying giving bortezomib together with dexamethasone, ifosfamide, carboplatin, and etoposide to see how well it works with or without rituximab in treating patients with relapsed or refractory AIDS-related non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and overall lymphoma response rate of bortezomib in combination with ifosfamide, carboplatin, and etoposide (ICE) with or without rituximab in patients with Epstein-Barr Virus (EBV)- and/or human herpes virus-8 (HHV-8)- positive relapsed or refractory HIV-associated non-Hodgkin lymphoma (NHL).

Secondary

* Evaluate the impact of bortezomib alone and in combination with rituximab) and ICE ([R] ICE) on serum HIV viral loads and APOBEC3G levels.
* Estimate the impact of bortezomib alone and in combination with (R)ICE on EBV and HHV-8 lytic activation using serum viral loads.
* Estimate the median response duration and 1 year overall survival rate of patients treated with this regimen.
* Evaluate the safety of bortezomib alone in patients with relapsed or refractory AIDS-associated lymphomas.
* Correlate EBV/HHV-8 viral load changes with lymphoma response.
* Compare the above outcomes to a parallel protocol employing ICE with or without rituximab in patients with EBV/HHV-8-negative AIDS-NHL to assess whether bortezomib has additional effects beyond (R)ICE alone.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib. Patients are assigned to 1 of 2 treatment groups.

* CD20-negative patients

  * Part A: Patients receive bortezomib IV over 3-5 seconds on days 1 and 8, dexamethasone IV and etoposide IV over 2 hours on days 8-10, and ifosfamide IV continuously over 24-hours and carboplatin IV over 2 hours on day 9. Treatment repeats every 28 days until the maximum tolerated dose (MTD) is determined. Patients who tolerate the MTD of bortezomib may move on to part B.
  * Part B: Patients receive bortezomib IV over 3-5 seconds at the MTD on days 1 and 8, dexamethasone IV on days 1-3 and 8, etoposide IV over 2 hours on days 1-3, and ifosfamide IV continuously over 24-hours and carboplatin IV over 2 hours on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Some patients may undergo hematopoietic stem cell transplantation (HSCT).
* CD20-positive patients

  * Part A: Patients receive bortezomib, dexamethasone, etoposide, ifosfamide, and carboplatin as in the CD20-negative patients part A group.
  * Part B: Patients receive rituximab IV on day 1. Patients also receive bortezomib, dexamethasone, etoposide, ifosfamide, and carboplatin as in the CD20-negative patients part B group. Some patients may undergo HSCT.

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for the effects of bortezomib on viral activation and replication via Taqman polymerase chain reaction (PCR), and for quantification of APOBEC3G levels via western blot. Similar studies are performed on the BCLB-1 EBV containing lines, as well as Daudi and other EBV-transformed B-lymphocyte lines via quantitative viral DNA PCR.

Patients complete the Functional Assessment of Cancer Therapy/GOG-Neurotoxicity Questionnaire, v4.0 at day 8 and week 4 of Part A and at least once per course of Part B for assessment of neuropathic pain and/or peripheral neuropathy.

After completion of study treatment, patients achieving complete response (CR) are followed at 2-4 weeks and then every 3 months for 1 year. Patients not achieving CR at completion of study treatment and declining further antineoplastic treatment are followed at 2-4 weeks and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed relapsed or refractory HIV-associated non-Hodgkin lymphoma (NHL)

  * Must have histologic or cytologic documentation of prior AIDS-associated NHL (i.e., at time of diagnosis) for clinically relapsed and/or refractory disease for which biopsy is not feasible
  * Must have documented HIV seropositivity
  * Must have documentation of Epstein-Barr Virus (EBV)- and/or human herpes virus-8 (HHV-8)- positive infection within the lymphoma (i.e., LMP-1, LANA expression, or positive Epstein-Barr-encoded RNAs [EBERs])

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 50-100%
* Life expectancy > 2 months
* ANC ≥ 1,000/mm³* (growth factor support allowed)
* Hemoglobin ≥ 8.0 g/dL* (growth factor support allowed)
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 mg/dL
* AST/ALT ≤ 2.5 times institutional upper limit of normal (ULN)
* Serum creatinine ≤ ULN
* Creatinine clearance ≥ 50 mL/min
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception NOTE: *Patients with lymphomatous involvement of the bone unable to meet hematologic criteria are allowed

Exclusion criteria:

* Peripheral neuropathy ≥ grade 2
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection

    * Opportunistic infections controlled by antimicrobial or suppressive therapy allowed, unless the investigator judges the infection likely to become life-threatening in the setting of multi-agent chemotherapy
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * NYHA class III or IV heat failure
  * Myocardial infarction within the past 6 months
  * Uncontrolled angina
  * Severe uncontrolled ventricular or other cardiac arrhythmias
  * Acute ischemia or active conduction system abnormalities by ECG
  * Serious psychiatric or medical illness, that would interfere with study compliance
* Social situations that would interfere with study compliance
* Acute active HIV-associated opportunistic infection requiring antibiotic treatment

  * Mycobacterium avium or candidiasis allowed unless concurrent therapy with moderate-to-strong CYP3A4 inducers or inhibitors is required
  * Chronic myelosuppressive agent therapy allowed provided hematologic criteria are met
* Hypersensitivity to compounds of similar chemical or biological composition to bortezomib, boron, mannitol, ifosfamide, carboplatin, or etoposide
* Concurrent malignancy except carcinoma in situ of the cervix, in situ anal cancer, nonmetastatic nonmelanoma skin cancer, or Kaposi's sarcoma not requiring systemic chemotherapy
* Active hepatitis B infection (hepatitis B surface antigen-positive), unless 1 of the following criteria are met:

  * Able to start dual anti-hepatitis B adefovir and telbivudine therapy prior to study
  * Receiving dual anti-hepatitis B therapy for at least 12 weeks prior to study with either agent active against HIV (i.e., entecavir, tenofovir, lamivudine, or emtricitabine)
* Concurrent grapefruit juice/fruit or green tea

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior adverse effects due to agents administered more than 3 weeks earlier
* Glucocorticoid therapy within the past 3 weeks allowed
* More than 3 weeks since prior chemotherapy
* More than 2 weeks since prior radiotherapy
* More than 14 days since prior and no other concurrent investigational agents (other than bortezomib)
* No concurrent moderate-to-strong CYP3A4 inducers or inhibitors other than protease inhibitors
* Concurrent stable (at least 12 weeks) antiretroviral regimen allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib | Assessed at end of cycle 1 for each group of 3 subjects
Overall lymphoma response rate | End of treatment
Safety as assessed using the CTCAE | Every cycle of treatment and all post-treatment visits

SECONDARY OUTCOMES:
Median overall survival at 1 year | 1 year post-treatment
Impact of bortezomib alone and in combination with rituximab, ifosfamide, carboplatin, and etoposide ([R]ICE) on serum HIV viral loads and APOBEC3G levels | baseline, day 2, 4, and 8 of week 1 of Part A, end of treatment
Impact of bortezomib alone and in combination with (R)ICE on EBV and HHV-8 lytic activation using serum viral loads | baseline, day 2, 4, and 8 of week 1 of Part A, end of treatment
Safety of bortezomib alone in patients with relapsed or refractory AIDS-associated lymphomas | Every cycle of treatment and all post-treatment visits
Correlation of EBV/HHV-8 viral load changes with lymphoma response | baseline, day 2, 4, and 8 of week 1 of Part A, end of treatment
Comparison of above outcomes to a parallel protocol employing ICE +/- rituximab in patients with EBV/HHV-8-negative AIDS-NHL to assess whether bortezomib has additional effects beyond (R)ICE alone | Upon availability of both studies' results

CONTACTS AND LOCATIONS:
Overall Officials: Erin G. Reid, MD, Study Chair — University of California, San Diego; William Wachsman, MD, Principal Investigator — University of California, San Diego
Locations (17):
- United States (17):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - University of California at Davis Center for Aids Research and Education Services, Sacramento, California
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Northwestern Cancer Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Pennsylvania Oncology Hematology Associates, Incorporated - Philadelphia, Philadelphia, Pennsylvania
  - Thomas Street Health Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Reid EG, Looney D, Maldarelli F, Noy A, Henry D, Aboulafia D, Ramos JC, Sparano J, Ambinder RF, Lee J, Cesarman E, Yahyaei S, Mitsuyasu R, Wachsman W; AIDS Malignancy Consortium. Safety and efficacy of an oncolytic viral strategy using bortezomib with ICE/R in relapsed/refractory HIV-positive lymphomas. Blood Adv. 2018 Dec 26;2(24):3618-3626. doi: 10.1182/bloodadvances.2018022095. PMID 30573564